CLINICAL TRIAL: NCT01582555
Title: Postoperative Nasal Irrigation Using Mucolytic Agents in Patients Undergoing Endoscopic Sinus Surgery
Brief Title: Postoperative Nasal Irrigation Using Mucolytic Agents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-12-AA-0089-CTIL
Record Dates: First submitted 2012-04-16; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Surgical Procedure, Unspecified
Keywords: mucolysis; QOL; endoscopy; sinus surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- saline irrigation (Experimental): a control arm (group A) of generic saline irrigation alone, irrigating with 20 mL per nostril tid for a total of 120 mL daily irrigation;
  Interventions: Drug: saline nasal irrigation alone
- intervention arm (group B), (Experimental): intervention arm (group B), which included generic N-Acetylcystine of 200 mg dissolved in 200 mL saline irrigated as per group A, 20 mL per nostril given tid daily (for a total of 120 mg).
  Interventions: Drug: dissolved N-Acetylcystine

INTERVENTIONS:
Drug: saline nasal irrigation alone — control arm (group A) of generic saline irrigation alone, irrigating with 20 mL per nostril tid for a total of 120 mL daily irrigation
  Other Names: Ocean, Saline Nasal Mist, Deep Sea Nasal Spray
  Arms: saline irrigation
Drug: dissolved N-Acetylcystine — intervention arm (group B), which included generic N-Acetylcystine of 200 mg dissolved in 200 mL saline irrigated as per group A, 20 mL per nostril given tid daily (for a total of 120 mg).
  Other Names: Ocean, Saline Nasal Mist, Deep Sea Nasal Spray
  Arms: intervention arm (group B),

SUMMARY:
Nasal irrigation techniques have been used for many years and been shown to improve symptoms of rhinosinusitis. Although there is a wealth of literature available, establishing treatment protocols can be difficult because of the great variability in recommended composition (seawater or hypertonic or isotonic saline with or without additives) and irrigation technique (variations in pressure and volume). Nasal irrigation is also used in many centers as part of postoperative treatment protocols and in particular has been recommended following endoscopic sinus surgery (ESS). Nasal crusting and thick nasal discharge have a negative impact on these patients quality of life (QOL). At the time of our study, there are no studies comparing irrigation with mucolysis with saline irrigation following ESS. The investigators aimed to assess whether mucolysis is effective at improving patients QOL and reducing postoperative signs as assessed endoscopically.

DETAILED DESCRIPTION:
The study will take place at Tel Aviv Sourasky medical center, otolaryngology outpatient clinic, a tertiary care academic hospital, for two years. It will be double-arm, open label, randomized controlled trial comparing two different methods of medical therapy following ESS. The allocation ratio is intended to be approximately equal for each arm. The two arms consisted of: a control arm (group A) of generic saline irrigation alone, irrigating with 20 mL per nostril tid for a total of 120 mL daily irrigation; and intervention arm (group B), which included generic N-Acetylcystine of 200 mg dissolved in 200 mL saline irrigated as per group A, 20 mL per nostril given tid daily (for a total of 120 mg). All medications will be used daily for the 3 months duration of the post-operative follow up. Patients will be instructed as to correct irrigation technique prior to discharge home from the hospital, and will be reminded of this technique at each postoperative clinic visit.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. Patient undergoing endoscopic sinus surgery

Exclusion Criteria:

1. Allergy to N-Acetylcysteine,
2. Any other nasal surgery performed concomitantly
3. Diagnosed with inflammatory (e.g. Wegener's granulomatosis, sarcoidosis) nasal pathology
4. Diagnosed with systemic conditions affecting the nose e.g. Cystic fibrosis, Kartagener's syndrome
5. Unable to give informed consent due to mental impairment
6. Unable to adhere follow up or treatment.
7. Patients requiring any additional nasal sprays (e.g. steroid sprays)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-06 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
change in QOL based on the Sino-Nasal Outcome Test-22 (SNOT-22) scores | 1 y
  The primary outcome measure is change in QOL based on the Sino-Nasal Outcome Test-22 (SNOT-22) scores.(5) SNOT-22 scores were chosen as the primary outcome due to the importance of studying patient QOL outcomes as opposed to imaging or endoscopy scores that often do not correlate with patients' subjective perceptions of disease severity.

SECONDARY OUTCOMES:
Lund-Kennedy endoscopic score (LKES) | 1y
  Secondary outcomes are the Lund-Kennedy endoscopic score (LKES) of each side of the nose that will be graded between 0 and 2 as recommended by the International Congress on Sinus Disease (Adhesions, Polyps, Crusting: 0 = none, 1 = middle meatus only, 2 = beyond middle meatus; Discharge: 0 = none, 1 = clear, thin, 2 = thick, purulent; Edema: 0 = none, 1 = mild, 2 = severe)

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Abergel, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel